CLINICAL TRIAL: NCT00746772
Title: Treatment of Oral Lichen Planus Lesions
Brief Title: Efficacy of Purslane in Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Qazvin university of medical sciences (school of dentistry), Qazvin university of medical sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 023
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Lichen Planus, Oral
Keywords: antioxidant; oral lichen planus; treatment; purslane
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Starch

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients with oral lichen planus
  Interventions: Drug: Purslane 235mg/day in one dosage
- 2 (Placebo Comparator): Patients with oral lichen planus
  Interventions: Drug: Placebo : one dosage

INTERVENTIONS:
Drug: Purslane 235mg/day in one dosage — Patients had been clinically with OLP and confirmed by histopathological findings were selected for the study. Gender, age, medical history, symptoms, types, size, and site of the lesions , duration of disease and other treatment used for this disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups .First group received systemic Purslane CAP with concentration antioxidant 235 mg/day in 1 dosage and second group used placebo CAP for 3 month. Each patients was examined at the beginning of the therapy ,and then 2 weeks after therapy and every 1 month up to 6 months
  Other Names: Portulaca oleracea.
  Arms: 1
Drug: Placebo : one dosage — Patients had been clinically with OLP and confirmed by histopathological findings were selected for the study. Gender, age, medical history, symptoms, types, size, and site of the lesions , duration of disease and other treatment used for this disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups .First group received systemic Purslane CAP with concentration antioxidant 235 mg/day in 1 dosage and second group used placebo CAP for 3 month. Each patients was examined at the beginning of the therapy ,and then 2 weeks after therapy and every 1 month up to 6 months .
  Other Names: starch
  Arms: 2

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory disease whose prevalence in the general population is 0.5 -2.2%.Oral lesions in OLP are chronic, rarely undergo spontaneous remission. Patients with OLP had significantly increased risk of oral squamous cell carcinoma, irrespective of the clinical type of OLP and therapy. there is currently no cure for OLP. Previous study demonstrated a decreased antioxidant defence and increased oxidative damage to lipids.DNA and proteins in lichen planus. This oxidative modifications point to pathophysiological alterations mainly within the basal cell layers of epidermis and at the dermoepidermal junction. Purslane is an excellent source of vitamin A,C and E and essential amino acids, has been described as a power food of the future because of its high nutritive and antioxidant properties. The purpose of the study was to determined the efficacy of Purslane in the treatment of oral lichen planus.

DETAILED DESCRIPTION:
Oral lichen planus is a chronic common inflammatory disorder affecting stratified squamous epithelia. The majority problem of OLP is development of oral squamous cell carcinoma , irrespective of the clinical type of OLP and therapy. Previous study demonstrated a decreased antioxidant defence and increased oxidative damage to lipids, DNA and proteins in lichen planus .This oxidative modifications point to pathophysiological alterations mainly within the basal cell layers of epidermis and at the dermoepidermal junction. So oxidative stress could be effective in pathogenesis of OLP. Purslane is an excellent source of vitamin A,C and E and essential amino acids, has been described as a power food of the future because of its high nutritive and antioxidant properties. Purslane also decreased the level of TNF-α and IL6, that are responsible for up-regulated adhesion molecules (in OLP lymphocyte T (T cell) recruited and retained in sub mucosa through receptors to endothelial adhesion molecule. and basal keratinocytes undergo apoptosis). The purpose of the study was to determined the efficacy of Purslane in the treatment of oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed symptomatic oral lichen planus: WHO histological criteria in combination with clinical appearance will be used for diagnosis
* Patients who had symptoms such as burning sensation, pain
* Patients not on any immunosuppressive or immunomodulatory treatment. In case they were,then such treatment should be stopped and a washout period of 1 month was given.
* Patients of both sexes between 30 to 70 year's old
* Patients who gave written informed consent
* Patients who were willing for evaluation in second week after therapy and every 1 month up to 6 months

Exclusion Criteria:

* The presence of histological signs of dysplasia
* Patients suffering from any localized or systemic disease
* Renal disease patients
* Pregnant patients
* Patients who can not continue the study for private or social reasons
* Patients who used lichenoid reaction including drugs

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Relief sign &symptom and clinical features | (every 1 month up to 6months)

SECONDARY OUTCOMES:
Relief sign &symptom and clinical features | (time frame6 months)

CONTACTS AND LOCATIONS:
Overall Officials: farzaneh aghahosseini, professor, Study Chair — Tehran University of Medical Sciences; farzaneh aghahosseini, professor, Study Director — Tehran University of Medical Sciences; hamidreza monsef esfehani, PHD, Study Director — Tehran University of Medical Sciences; Katayun Borhanmojabi, DDS-MS, Study Director — Qazvin University Of Medical Sciences; Shahroo Etemad moghadam, DDS-MS, Study Director — Qazvin University Of Medical Sciences; Aida(touba) Karagah, DDS, Principal Investigator — Qazvin University Of Medical Sciences; Eraj mirzaii, physiology, Study Director — Tehran University of Medical Sciences
Locations (1):
- Qazvin university of medical sciences, Qazvin, Qazvin Province, Iran